CLINICAL TRIAL: NCT06128499
Title: Development a Core Set for Adults With Cystic Fibrosis Based on the International Classification of Functioning, Disability, and Health (ICF)
Brief Title: Development a Core Set for Adults With Cystic Fibrosis Based on the ICF
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nisa Akyazı, B.Sc., Principal Investigator, Hacettepe University
Other Study IDs: GO 23/58
Record Dates: First submitted 2023-05-03; First posted 2023-11-13 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; ICF; ICF Core Set
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic Fibrosis (CF) affects more than one body system, mainly respiratory and digestive.The quality of life of individuals with CF is adversely affected by the increasing treatment burden in addition to multi-system involvement. The International Classification of Functioning, Disability and Health (ICF) describes human functioning and states of disability and provides a framework for organizing this information. ICF Core Sets are created by selecting the appropriate categories for the current disease from the ICF classification. ICF Core Sets are smaller than ICF, allowing practical evaluation based on ICF in clinical use. It evaluates the current situation of the patient quickly and practically, and improves interdisciplinary cooperation. Our study, it was aimed to develop a core set that quickly and practically evaluates the current state of the patient with CF in Turkey, based on ICF, and increases coordination within the interdisciplinary team.

In our study, the established, very comprehensive, scientific and evidence-based guide that should be followed while creating the ICF core set will be followed. The guide consists of 4 stages: The first stage is the literature review which allows us to see the disease from the perspective of the researcher by scanning the studies on CF in the last 10 years. The second stage is the patient interview, which includes interviewing these individuals, and allows us to see the disease from the perspective of individuals diagnosed with CF. The third phase is the expert questionnaire, which we will look at from the perspective of health professionals who are knowledgeable about treating individuals with CF. The fourth stage is the consensus stage, where the final core set is decided, which includes team discussion. With the final core set developed as a result of these stages, a core set that will quickly and practically evaluate the current situation of the patient with CF in Turkey based on ICF and increase coordination within the interdisciplinary team will be ensured.

Hypothesis(s) and purpose(s) on which this thesis proposal is based:

H1: The ICF Core Set will be instrumental in understanding CF-specific health, disability, and function.

H2: It will be a step in the development of a standard tool for the assessment of adults with CF.

In our study, we propose to examine CF from the perspective of the researcher as a result of the literature review, from the perspective of the patient as a result of the qualitative research, from the perspective of the health professional as a result of the expert survey, to create a core set specific to these patients, and thus to see the different characteristics of individuals with CF in terms of function, activity, participation, and environmental factors.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a chronic, progressive, and autosomal recessive disease that shortens life expectancy caused by mutations in the Cystic Fibrosis Transmembrane Regulator (CFTR ) gene. It affects more than one body system, mainly the respiratory and digestive. The quality of life of individuals with CF is adversely affected by the increasing treatment burden in addition to multi-system involvement. Disorders in CF affect the structures and functions of various systems, especially the respiratory and digestive systems. This influence causes a decrease in the activity and participation of individuals with CF. Factors such as age, gender, and coping strategies of individuals may affect the severity of these symptoms in individuals with CF. Scientific advances in biology in CF have provided therapeutic diversity, thereby improving patient care and prolonging survival. Pancreatic enzyme supplementation, airway cleansing, long-term antimicrobial therapy for respiratory tract infection, and nutritional supplements are among the current treatments. CFTR modulators, which have been developed in recent years to improve CFTR protein function, have been reported to greatly benefit individuals with CF. It can be said that the life expectancy of individuals with CF is prolonged by developing-changing treatment strategies and multidisciplinary approaches. It has been reported in international records that approximately 150,000 patients worldwide have been diagnosed with CF. The incidence of the disease is estimated to be 1/3,000 live births in Northern Europe, 1/4.000-10,000 in Latin Americans, and 1/15,000-20,000 in African-Americans. There is limited number of studies on the incidence of CF in Turkey. In the study conducted by Gurson in 1973, the incidence of CF was determined as 1/3,000. According to the annual records of the Cystic Fibrosis Society of Turkey, there are 1930 CF patients followed in various centers in 2021 in Turkey. The International Classification of Functioning, Disability, and Health (ICF) describes human functioning and states of disability and provides a framework for organizing this information. The World Health Organization approved the ICF in 2001 to classify and describe patients' functions within the specific social and environmental context in which they live.

ICF not only defines the health status of individuals but also allows health professionals to create a common language. The ICF includes five interrelated components: body functions (b), body structures (s), activity and participation (d), environmental factors (e), and personal factors. ICF, each of these components is hierarchically structured for one, followed by the second, third, and fourth levels. As you progress from the first to the fourth level, the descriptions of the categories become more detailed. Since it contains ICF 1495 categories, it is practically difficult to apply in clinical settings. Disease-specific assessment tools are required because diseases affect people in many ways. Therefore, there is a need to create disease-specific subsets of ICF categories that will make it easier to apply in the clinic. For this reason, the ICF Core Set is designed to be purposeful, and essential and can be used in daily clinical practice. ICF Core Sets are created by selecting the appropriate categories for the current disease from the ICF classification. ICF Core Sets are smaller than ICF, allowing practical evaluation based on ICF in clinical use. It evaluates the current situation of the patient quickly and practically, and improves interdisciplinary cooperation.Work is underway to develop the ICF Core Set, which is internationally recognized shortlist of the most relevant and essential ICF categories that can be used to assess and document the condition of patients living with a particular health condition. Core sets have been developed for various health conditions such as neurological, pediatric, cardiopulmonary, musculoskeletal, and cancer. Studies investigating Cystic Fibrosis from the ICF perspective are limited, but there are no studies within the scope of the core set. Our study, it was aimed to develop a core set that quickly and practically evaluates the current situation of the patient with CF in Turkey based on ICF and increases the coordination within the interdisciplinary team.

In our practice, we will follow an established, very comprehensive, scientific and evidence-based guide published by the 'ICF Research Branch', which should be followed when creating the ICF-Core Set. The research consists of 4 steps.

A 'literature review' that allows us to view primary care CF from the perspective of the investigator. In this step, studies on CF for the last 10 years will be searched from various databases (PUBMED, Scopus, Embase).

Literature Review-Inclusion Criteria

* Studies with individuals over the age of 18 with a diagnosis of Cystic Fibrosis
* Studies published in the last 10 years
* Studies in English
* Randomized controlled, clinical control study, observational studies, cross-sectional studies, qualitative studies

Literature Review - Exclusion Criteria

-Psychometric and prevention studies, phase II clinical research studies, studies with laboratory parameters only, animal experiments, letters, comments and editorials

Qualitative research that allows us to view second-line CF from the perspective of individuals diagnosed with CF. It is planned to reach adult individuals who are followed up with the diagnosis of CF in Hacettepe University Department of Chest Diseases and referred to Hacettepe University Faculty of Physical Therapy and Rehabilitation. Focus group discussions with a maximum of 7 people will be held. With the guidance of the moderator, 6 open-ended questions covering the components of the ICF will be asked.

Qualitative Research- Inclusion Criteria

* Individuals over the age of 18 with a diagnosis of CF
* Volunteering to participate in research

The 'expert survey' allows us to see tertiary CF through the eyes of healthcare professionals. At this step, 6 open-ended questions covering ICF components for individuals with CF will be asked via e-mail to healthcare professionals who treat individuals with CF or have experience in research in this field. We are planning to reach the physicians working in the field of CF in the Hacettepe University Chest Diseases Department and the people with whom these physicians are in the National Cystic Fibrosis Patient Registry and collaborate. We plan to reach physiotherapists who work with patients diagnosed with CF academically and clinically at Hacettepe University Faculty of Physical Therapy and Rehabilitation, and physiotherapists who have experience in this field in different centers. Other health professionals (dieticians, nurse) who are familiar with the problems related to CF will be reached with the cooperation of physicians and physiotherapists.

Expert Questionnaire-Inclusion Criteria

* Have at least three months of experience in treating and/or researching individuals with CF, with knowledge of CF-related problems
* Volunteering to participate in research

The fourth step is the 'consensus' that we will create the final Core Set as a result of the data we collect. A multidisciplinary team (Physician, Physiotherapist, Dietitian, Nurse) meeting will be held for the Short Core Set created in this step.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 with a diagnosis of CF
* Volunteering to participate in research

Exclusion Criteria

* Not volunteering to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to reach adult individuals who are followed up with the diagnosis of CF in the Hacettepe University Department of Chest Diseases and referred to the Hacettepe University Faculty of Physical Therapy and Rehabilitation. Focus group discussions with a maximum of 7 people will be held. With the guidance of the moderator, 6 open-ended questions covering the components of the ICF will be asked.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Literature Review | 08.05.23- 01.12.23
  A 'literature review' that allows us to view primary care CF from the perspective of the investigator. In this step, studies on CF for the last 10 years will be searched from various databases (PUBMED, Scopus, Embase).

SECONDARY OUTCOMES:
Qualitative Research | 08.05.23- 01.12.23
  Qualitative research allows us to see from the perspective of individuals diagnosed with CF through a questionnaire.

OTHER OUTCOMES:
Expert Survey | 08.05.23- 01.12.23
  6 open-ended questions covering ICF components for individuals with CF will be asked via e-mail to healthcare professionals who treat individuals with CF or have experience in research in this field

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shteinberg M, Haq IJ, Polineni D, Davies JC. Cystic fibrosis. Lancet. 2021 Jun 5;397(10290):2195-2211. doi: 10.1016/S0140-6736(20)32542-3. PMID 34090606
- [Background] Mandrusiak A, MacDonald J, Watter P. The International Classification of Functioning, Disability and Health: an effective model for describing young people with cystic fibrosis. Child Care Health Dev. 2009 Jan;35(1):2-4. doi: 10.1111/j.1365-2214.2008.00903.x. No abstract available. PMID 19522999
- [Background] Lopes-Pacheco M. CFTR Modulators: The Changing Face of Cystic Fibrosis in the Era of Precision Medicine. Front Pharmacol. 2020 Feb 21;10:1662. doi: 10.3389/fphar.2019.01662. eCollection 2019. PMID 32153386
- [Background] Kerem B, Rommens JM, Buchanan JA, Markiewicz D, Cox TK, Chakravarti A, Buchwald M, Tsui LC. Identification of the cystic fibrosis gene: genetic analysis. Science. 1989 Sep 8;245(4922):1073-80. doi: 10.1126/science.2570460.
- [Background] O'Sullivan BP, Freedman SD. Cystic fibrosis. Lancet. 2009 May 30;373(9678):1891-904. doi: 10.1016/S0140-6736(09)60327-5. Epub 2009 May 4. PMID 19403164
- [Background] Gurson CT, Sertel H, Gurkan M, Pala S. Newborn screening for cystic fibrosis with the chloride electrode and neutron activation analysis. Helv Paediatr Acta. 1973 May;28(2):165-74. No abstract available. PMID 4706142
- [Background] 7.https://www.kistikfibrozisturkiye.org/wp-content/uploads/2022/11/UKKS-2021-raporu-2.pdf
- [Background] Kabakçı E, and Gogus A 2004 International classification of functioning, disability and health Ankara:Başbakanlık Özürlüler İdaresi Başkanlığı
- [Background] Rauch A, Cieza A, Stucki G. How to apply the International Classification of Functioning, Disability and Health (ICF) for rehabilitation management in clinical practice. Eur J Phys Rehabil Med. 2008 Sep;44(3):329-42. PMID 18762742
- [Background] Yen TH, Liou TH, Chang KH, Wu NN, Chou LC, Chen HC. Systematic review of ICF core set from 2001 to 2012. Disabil Rehabil. 2014;36(3):177-84. doi: 10.3109/09638288.2013.782359. Epub 2013 May 7. PMID 23651126
- [Background] ICF Research Branch - ICF Core Sets Projects. https://www.icf-research-branch.org/icf-core-sets-projects2 (accessed November 30, 2022)
- [Background] Coenen M, Cieza A, Freeman J, Khan F, Miller D, Weise A, Kesselring J; Members of the Consensus Conference. The development of ICF Core Sets for multiple sclerosis: results of the International Consensus Conference. J Neurol. 2011 Aug;258(8):1477-88. doi: 10.1007/s00415-011-5963-7. Epub 2011 Mar 4. PMID 21373900
- [Background] Cieza A, Kirchberger I, Biering-Sorensen F, Baumberger M, Charlifue S, Post MW, Campbell R, Kovindha A, Ring H, Sinnott A, Kostanjsek N, Stucki G. ICF Core Sets for individuals with spinal cord injury in the long-term context. Spinal Cord. 2010 Apr;48(4):305-12. doi: 10.1038/sc.2009.183. Epub 2010 Jan 12. PMID 20065984
- [Background] Schiariti V, Masse LC, Cieza A, Klassen AF, Sauve K, Armstrong R, O'Donnell M. Toward the development of the International Classification of Functioning Core Sets for children with cerebral palsy: a global expert survey. J Child Neurol. 2014 May;29(5):582-91. doi: 10.1177/0883073813475481. Epub 2013 Feb 21. PMID 23435282
- [Background] Boldt C, Grill E, Wildner M, Portenier L, Wilke S, Stucki G, Kostanjsek N, Quittan M. ICF Core Set for patients with cardiopulmonary conditions in the acute hospital. Disabil Rehabil. 2005 Apr 8-22;27(7-8):375-80. doi: 10.1080/09638280400013982. PMID 16040539
- [Background] Boonen A, Braun J, van der Horst Bruinsma IE, Huang F, Maksymowych W, Kostanjsek N, Cieza A, Stucki G, van der Heijde D. ASAS/WHO ICF Core Sets for ankylosing spondylitis (AS): how to classify the impact of AS on functioning and health. Ann Rheum Dis. 2010 Jan;69(1):102-7. doi: 10.1136/ard.2008.104117. PMID 19282309
- [Background] Tschiesner U, Rogers S, Dietz A, Yueh B, Cieza A. Development of ICF core sets for head and neck cancer. Head Neck. 2010 Feb;32(2):210-20. doi: 10.1002/hed.21172. PMID 19572286
- [Background] Bagci R, Vardar-Yagli N, Saglam M, Calik Kutukcu E, Inal-Ince D, Sener F, Damadoglu E. Body functions and structure, activity, and participation limitations of adult cystic fibrosis patients under the international classification of functioning, disability, and health framework. Physiother Theory Pract. 2023 Jul 3;39(7):1417-1427. doi: 10.1080/09593985.2022.2041780. Epub 2022 Feb 22. PMID 35192420
- [Background] McLeod C, Smyth AR, Messer M, Schultz A, Wood J, Norman R, Blyth CC, Webb S, Elliott Z, Van Devanter D, Stephenson AL, Tong A, Snelling TL. Protocol for establishing a core outcome set for evaluation in studies of pulmonary exacerbations in people with cystic fibrosis. BMJ Open. 2022 Sep 23;12(9):e056528. doi: 10.1136/bmjopen-2021-056528. PMID 36153014
- [Background] Selb M, Escorpizo R, Kostanjsek N, Stucki G, Ustun B, Cieza A. A guide on how to develop an International Classification of Functioning, Disability and Health Core Set. Eur J Phys Rehabil Med. 2015 Feb;51(1):105-17. Epub 2014 Apr 1. PMID 24686893
- [Background] Cieza A, Geyh S, Chatterji S, Kostanjsek N, Ustun B, Stucki G. ICF linking rules: an update based on lessons learned. J Rehabil Med. 2005 Jul;37(4):212-8. doi: 10.1080/16501970510040263. PMID 16024476
- See also: National Cystic Fibrosis Registry (TÜRKİYE) — https://www.kistikfibrozisturkiye.org/wp-content/uploads/2022/11/UKKS-2021-raporu-2.pdf
- See also: icf-research-branch — https://www.icf-research-branch.org/icf-core-sets-projects2